CLINICAL TRIAL: NCT03890796
Title: Application of Activity Scheduling to Enhance Quality of Life for Older Adults With Dementia
Brief Title: Activity Scheduling for Older Adults With Dementia
Acronym: AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Frank LAI, Principal Investigator, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSEARS20190322004
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Older Adults With Mild to Moderate Level of Dementia

STUDY DESIGN:
Intervention Model Description: The study model is longitudinal, single-blind, parallel group experiment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors were blinded regarding the participants' belonging to the two study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dementia Care Education and Activity Scheduling Group (DE&AS) (Experimental): Will received both dementia care education and activity scheduling
  Interventions: Behavioral: Activity Scheduling; Behavioral: Educational
- Dementia Care Education Group (DE) (Sham Comparator): Will received dementia care education
  Interventions: Behavioral: Educational

INTERVENTIONS:
Behavioral: Activity Scheduling — AS is strategy for behavioral activation that has also been used with success in people with dementia, after the training of their caregivers. A certified occupational therapist will train up the caregivers of dementia in conducting AS activities for participants in experimental group
  Other Names: Experimental
  Arms: Dementia Care Education and Activity Scheduling Group (DE&AS)
Behavioral: Educational — A serial of dementia care education program with a weekly theme of topics like: importance of exercise and healthy eating, sleep management, counselling, acceptance therapy, commitment therapy, reminiscence therapy.
  Other Names: Control

SUMMARY:
This study is to evaluate the results from an intervention designed to encourage older adults with dementia for their engagement in activities through their active participation of activity scheduling (AS).

DETAILED DESCRIPTION:
The study compares two interventions by using a 12-week longitudinal randomized controlled trial. For the first 2 weeks, all participants receive the same health care education program. Then for the following 10 weeks, participants will be randomized to either one of the two following groups with different conditions. For the control group, participants receive ten session of dementia care education. For the experimental activity scheduling group, participants receive ten session of dementia care education, plus weekly activity scheduling (AS) practice that focus on pleasant event scheduling and improving communication.

ELIGIBILITY:
Inclusion Criteria:

* patients had to have an age of at least 65 years,
* a diagnosis for dementia in medical history and had to meet international classification of disease-10 criteria for dementia,
* diagnosed by a psychiatrist.
* patients had to have cognitive impairment, as determined by the Montreal Cognitive Assessment

Exclusion Criteria:

* any major neurological illness other than AD,
* any psychiatric disorder or a known history of substance abuse.

Ages: 65 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the Caregiver Burden Interview Scale (Chinese ZBIS) | 12 months
  This is a 22-item instrument measures caregiver stress. Areas assessed include the perceived health and psychological well-being of the caregiver, financial impact, social life, and the relationship between the caregiver and the care recipient. The Chinese version has been tested with family caregivers of community-dwelling persons with dementia. Its correlation with the General Health Questionnaire (GHQ) was 0.59 (p<0.001). The intraclass correlation coefficient was 0.99. The split-half correlation coefficient was 0.81 (Chan, 2005). higher values represent higher stress level of caregivers

SECONDARY OUTCOMES:
Revised Memory and Behavior Problem Checklist (RMBPT) | 12 months
  24-item questionnaire to assess three domains of problematic behaviors in older adults
Chinese Caregiver Activity Survey (Chinese CAS) | 12 months
  The 6-item CAS to assess the amount of time that caregivers spend taking care of people with dementia during the 24 hours before the investigation. It covers six areas of daily living: communication, using transportation, dressing, eating, looking after the appearance of people with dementia, and supervising them. The total score the Chinese CAS is calculated by summing the total time that caregivers spend on assistance with these areas of daily living (Prince, 2004).

OTHER OUTCOMES:
Cantonese Chinese version of Quality of Life in Chinese Alzheimer's Disease (The Cantonese Chinese QOL-AD) | 12 months
  13 items to measure QoL of participants. higher values represent a better QoL. outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Welfare Club Western District, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen CK, Wittrup-Jensen KU, Lolk A, Andersen K, Kragh-Sorensen P. Ability to perform activities of daily living is the main factor affecting quality of life in patients with dementia. Health Qual Life Outcomes. 2004 Sep 21;2:52. doi: 10.1186/1477-7525-2-52. PMID 15383148
- [Background] Dozeman E, van Schaik DJ, van Marwijk HW, Stek ML, Beekman AT, van der Horst HE. Feasibility and effectiveness of activity-scheduling as a guided self-help intervention for the prevention of depression and anxiety in residents in homes for the elderly: a pragmatic randomized controlled trial. Int Psychogeriatr. 2011 Aug;23(6):969-78. doi: 10.1017/S1041610211000202. Epub 2011 Feb 22. PMID 21338550